CLINICAL TRIAL: NCT07207733
Title: Feasibility Study of PcyCare (Pregnancy Care) : A Self-Learning Educational Platform for Pregnant Women
Acronym: PcyCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurul Jannah, M.Tr.Keb (Other)
Collaborators: Lincoln University College Malaysia (Other)
Responsible Party: Sponsor-Investigator, Nurul Jannah, M.Tr.Keb, Feasibility Study of PcyCare (Pregnancy Care) : A Self-Learning Educational Platform for Pregnant Women, Lincoln University College
Organization: Lincoln University College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LUC20230708005; LUC20230708005 (Other: Lincoln University College Malaysia)
Record Dates: First submitted 2025-09-11; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy
Keywords: Pregnancy care; Prenatal education; Self-learning platform; Feasibility study; Digital health intervention

STUDY DESIGN:
Intervention Model Description: Participants will use the PcyCare self-learning educational platform for one week. There is no randomization, crossover, or control group. The study aims to evaluate the feasibility, usability, and content quality of the platform based on feedback from pregnant women as primary users and expert reviewers, including maternal health specialists and IT/media experts.
Masking Description: Not applicable. This study does not involve masking or blinding as all participants and expert reviewers are aware of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PcyCare (Pregnancy Care) Users (Experimental): Participants in this arm, consisting of pregnant women, used the PcyCare self-directed education platform for one week. Participants accessed educational modules covering nutrition, pregnancy warning signs, mental health, and childbirth preparation. This intervention included interactive content, instructional videos, and quizzes. Data on ease of use, participant satisfaction, and increased understanding were collected through questionnaires. In addition, input from expert assessors in the fields of obstetrics and information technology will be used to assess the quality of the content and the suitability of the platform.
  Interventions: Device: PcyCare: Self-Directed Education Platform for Pregnant Women

INTERVENTIONS:
Device: PcyCare: Self-Directed Education Platform for Pregnant Women — This intervention involves the use of the PcyCare self-directed education platform by pregnant women for one week. Participants will access educational modules on nutrition, pregnancy warning signs, mental health, and childbirth preparation. The platform includes interactive content, instructional videos, and quizzes to enhance participants' understanding. Data on ease of use, satisfaction, and increased understanding will be collected through questionnaires. In addition, midwives/practicing midwives and information technology/media experts will assess the quality of the platform's content and features through expert reviews to evaluate the platform's suitability and improvements before wider trials.
  Other Names: PcyCare Self-Learning Educational Platform; Digital Pregnancy Care Platform

SUMMARY:
Brief Summary - PcyCare (Pregnancy Care Aplication) (with expert participants)

Objective:

This study aims to evaluate the feasibility and usefulness of the PcyCare self-directed education platform for pregnant women. This platform provides information on nutrition, pregnancy warning signs, mental health, and childbirth preparation.

Key questions:

Is PcyCare easy to use for pregnant women? Do the platform's materials and features help improve participants' understanding of pregnancy and childbirth? How do subject matter experts and information technology experts assess the quality of the platform's content and features?

Procedure:

Pregnant women will use PcyCare for one week, accessing educational materials, watching videos, and completing interactive quizzes. Their understanding and experience will be evaluated through feasibility and satisfaction questionnaires.

Content experts (midwifery lecturers/practicing midwives) and media/IT experts will assess the suitability of the platform's content and features through expert reviews and provide suggestions for improvement.

Expected results:

Information about ease of use, content quality, effectiveness of interactive features, and input from experts to refine the platform before wider trials.

DETAILED DESCRIPTION:
Detailed Description The PcyCare platform was developed as a self-directed educational medium for pregnant women, with the aim of improving understanding of nutrition, pregnancy warning signs, mental health, and childbirth preparation. This study aims to evaluate the feasibility, ease of use, and content quality of the platform prior to wider implementation, while also obtaining input from experts for platform refinement.

This study involved 10 pregnant women as primary users. During the one-week study period, participants accessed the platform via smartphone or computer, read educational materials, watched interactive videos, and completed quizzes. Researchers collected data through feasibility and satisfaction questionnaires and assessed participants' understanding before and after using the platform. This activity aimed to determine whether the platform was easy to use and could improve pregnant women's understanding.

In addition, the study also involved 8 subject matter experts (midwifery lecturers/practicing midwives) and 5 information technology/media experts as evaluators of the platform's content and features. The experts assessed the scientific accuracy, completeness of the material, language, cultural appropriateness, visual quality, and interactivity of the platform using a special assessment instrument (expert review). Input from experts will be used to improve and refine the platform before it is tested more widely.

The results of the study are expected to provide information on ease of use, content quality, effectiveness of interactive features, and recommendations for improvement from experts. This study will serve as a basis for improving the feasibility and quality of PcyCare, so that the platform can be used as an effective and safe self-education medium for pregnant women at various educational and socio-cultural levels.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 20-35 years
* Gestational age between 12 and 36 weeks
* Able to read and understand the language used in the PcyCare platform
* Owns a smartphone, tablet, or computer with internet access
* Provides informed consent to participate

Exclusion Criteria:

* High-risk pregnancy requiring intensive medical care
* Severe psychiatric or cognitive disorders that would prevent platform use
* Participation in another conflicting educational or intervention study

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Women (Female)
Enrollment: 10 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Usability of PcyCare Platform by Pregnant Women assessed using a Custom User Experience Questionnaire | 1 weeks after initial use of the PcyCare platform
  The assessment evaluated PcyCare platform usability by pregnant women using a 30-item feasibility questionnaire across six dimensions: navigation, interactivity, material accessibility, comfort, usefulness, and overall satisfaction. The form covered respondent identity and quantitative ratings on a 4-point Likert scale (1=Not appropriate to 4=Very appropriate). Scores ranged from 30-120, with feasibility defined as ≥3.00 (Feasible), 2.50-2.99 (Conditionally Feasible), and <2.50 (Not Feasible). Ten pregnant women participated. Results showed strong validity: 22 items scored I-CVI=1.00, 8 items I-CVI=0.75, yielding S-CVI=0.93. This indicates the instrument demonstrates high content validity and effectively measures user experiences and platform feasibility.

SECONDARY OUTCOMES:
Content Quality Evaluation of PcyCare Platform by Subject Matter Experts using Content Validity Index (CVI) | Performed immediately after the platform is tested by experts (1 week)
  The content quality of the PcyCare platform was evaluated using a 28-item questionnaire completed by 8 subject matter experts. The items covered ten key aspects: scientific accuracy, content completeness, language clarity, cultural and local relevance, visual/media support, interactivity and self-learning, timeliness and consistency, practical usefulness, information safety, and overall evaluation. Each item was rated on a 4-point Likert scale (1=Not Relevant to 4=Highly Relevant), with scores ranging from 28-112. Feasibility was interpreted as ≥3.00 (Feasible), 2.50-2.99 (Conditionally Feasible), and <2.50 (Not Feasible). Results showed strong validity: 21 items had I-CVI=1.00, 7 items had I-CVI=0.75, and the S-CVI was 0.94, confirming excellent overall content validity of the expert assessment instrument.

OTHER OUTCOMES:
Technical Feasibility and Media Quality Evaluation by Information Technology and Media Experts using Structured Expert Review Questionnaire | 1 Week
  The technical feasibility and media quality of the PcyCare platform were evaluated using a 28-item questionnaire reviewed by 5 IT and media experts. The items covered 10 aspects: scientific accuracy, content completeness, language clarity, cultural relevance, visual/media support, interactivity, timeliness and consistency, practical usefulness, information safety, and overall evaluation. Each item was rated on a 4-point Likert scale (1=Not Relevant to 4=Highly Relevant), with scores ranging from 28-112. Feasibility was defined as ≥3.00 (Feasible), 2.50-2.99 (Conditionally Feasible), and <2.50 (Not Feasible). Results showed strong validity: 24 items had I-CVI=1.00, 4 items had I-CVI=0.75, with S-CVI=0.96, confirming excellent overall content validity of the expert review instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Nurul Jannah, M.Tr.Keb, Principal Investigator — Lincoln University College Malaysia
Locations (1):
- Disctrict, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared outside the research team to protect the privacy and confidentiality of pregnant participants. Data contain sensitive personal health information, and sharing it could risk participant identification. Any future decision to share data will comply with applicable privacy regulations and ethical guidelines.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT07207733/Prot_SAP_ICF_000.pdf